CLINICAL TRIAL: NCT04086849
Title: Analysis of Patterns of Recurrence in Head and Neck Cancer Using Clinicopathomic Markers
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. William Tran, Radiation Therapist Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 087-2019
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Neoplasm; Squamous Cell Carcinoma of Head and Neck
Keywords: radiomics; pathomics; head and neck cancer; biomarkers; machine learning; artificial intelligence; squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fixed tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radiomic, pathomic, and clinical markers — This is a non-interventional study.

SUMMARY:
Here, the investigators will develop a clinicopathomic assay from biomarkers obtained from digital pathologies of resected whole-mount oral cavity and oropharyngeal squamous cell carcinoma (OCSCC and OPSCC) specimens with the goal of administering personalized novel image-guided therapies immediately after primary surgical management in OCSCC and OPSCC patients. The primary aim is to determine the association between clinicopathomic biomarkers and LRR. The secondary aim is to develop a clinicopathomic risk score (assay) such that a decision-support tool can be used by physicians for measuring the benefit of additional therapies (i.e. conventional chemotherapy +/- radiation or administering dose-escalated chemoradiation) in the adjuvant setting to reduce LRR rates.

DETAILED DESCRIPTION:
The proposed study is significant for developing personalized treatments. The proposed research will yield high rewards to patients by providing additional information to clinicians for better prognostication and potentially adapting adjuvant treatments to improve the survival of patients with OCSCC or OPSCC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be men and women age 18+
* Confirmed diagnosis of oral cavity or oropharyngeal squamous cell carcinoma
* Participants must have received or will undergo surgery to excise the primary oropharyngeal tumor.

Exclusion Criteria:

* Participants who had other primary cancers prior to oral cavity or oropharyngeal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll women and men with a pathologically-confirmed diagnosis of early-stage oral cavity or oropharyngeal squamous cell carcinoma that undergo surgery to excise the tumor.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Time to locoregional recurrence | Up to 60 months
  Evaluating the time until a recurrence event has occurred in the oral cavity or oropharyngeal region

SECONDARY OUTCOMES:
Time to distant metastasis | Up to 60 months
  Evaluating onset of distant metastasis
Time to death | Up to 60 months
  Evaluating time to cancer-related death

CONTACTS AND LOCATIONS:
Overall Officials: William Tran, MRT(T), PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized. Digital pathology images and anonymized clinical data will be deposited into the National Cancer Institute (NCI) data sharing repository, including The Cancer Imaging Archive (TCIA). Digital pathology images will also be annotated to facilitate analysis for other investigators. Computational methods, source-codes and instructions will be deposited to the open-source coding repository, GitHub (www.github.com).
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Digital pathology images, anonymized clinical data, source codes, and computational methods will be deposited to open-source repositories.